CLINICAL TRIAL: NCT03875937
Title: Pharmacokinetics of Intramuscular Tranexamic Acid in Trauma Patients: a Clinical Trial
Brief Title: The Trauma INtramuscular Tranexamic Acid Clinical Trial
Acronym: TraumaINTACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Barts & The London NHS Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); University of Versailles (Other); JP Moulton Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019/KEP/218; 2019-000898-23 (EudraCT Number)
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-02

CONDITIONS: Traumatic Haemorrhage
Keywords: tranexamic acid; pharmacokinetic; intramuscular

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, multicentre, pharmacokinetic study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tranexamic acid 1 gram intramuscularly (Experimental): Patients will receive a 1 gram dose of TXA by IM injection at least 1 hour and 30 minutes after their initial IV injection received at the scene or on arrival to hospital. The IM dose will be given as two 5mL (0.5 gram each) injections into the thigh (rectus femoris or vastus lateralis), gluteal or deltoid muscles, depending on the clinical scenario (e.g. taking into account the type of injury). Injections should be given in a non-injured muscle.
  Interventions: Drug: Tranexamic 1 gram

INTERVENTIONS:
Drug: Tranexamic 1 gram — To be administered intramuscularly (2 injections)

SUMMARY:
Intramuscular injection of tranexamic acid (TXA) would increase its use in situations where administration of intravenous drugs is difficult. The investigators aim to assess the population pharmacokinetics of intramuscular TXA in trauma patients.

Primary endpoint: Serum TXA concentrations over time. Secondary endpoints: Local reactions at injection sites and adverse events

DETAILED DESCRIPTION:
A prospective, open-label, multicentre, pharmacokinetic study conducted in the UK hospital. Potential eligible patients will have received a 1 gram IV dose of TXA at the scene of the injury or on arrival in hospital and a second dose is clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Adult (appear to be at least 16 years old) trauma patients who have received 1 gram of intravenous TXA for the management of haemorrhage in whom a second dose is clinically indicated are eligible.

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Concentration of serum TXA concentrations over time. | Blood samples will be taken pre-dose and up to 11 hours after IM TXA

SECONDARY OUTCOMES:
Number of participants with Injection sites reactions | death, discharge or day seven (whichever comes first)
Number of adverse events reported by type | death, discharge or day 7 (whichever comes first)
  adverse events will be coded using MedDRA

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur-Still, Principal Investigator — London School of Hygiene and Tropical Medicine; Ian Roberts, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- United Kingdom (2):
  - The Royal London Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Dataset used for main analysis will be made freely available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: freely available 1 year after main publication
Access Criteria: Free login to website required for monitoring usage of data
URL: https://freebird.lshtm.ac.uk

REFERENCES:
- [Derived] Grassin-Delyle S, Shakur-Still H, Picetti R, Frimley L, Jarman H, Davenport R, McGuinness W, Moss P, Pott J, Tai N, Lamy E, Urien S, Prowse D, Thayne A, Gilliam C, Pynn H, Roberts I. Pharmacokinetics of intramuscular tranexamic acid in bleeding trauma patients: a clinical trial. Br J Anaesth. 2021 Jan;126(1):201-209. doi: 10.1016/j.bja.2020.07.058. Epub 2020 Sep 30. PMID 33010927